CLINICAL TRIAL: NCT01849900
Title: Efficacy Study of the Preconception Reproductive Knowledge Promotion Intervention
Brief Title: Preconception Reproductive Knowledge Promotion (PREKNOP)
Acronym: PREKNOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Calvin College (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Adejoke Ayoola, Dr., Calvin College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 70315
Record Dates: First submitted 2013-05-01; First posted 2013-05-09 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Pregnancy
Keywords: Menstrual cycle; Ovulation time; pregnancy recognition; Community-based participatory research; Unintended pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Lifestyle (Other): 60 women randomly assigned to the control group
  Interventions: Behavioral: Healthy Lifestyle
- Knowing your body (Other): 60 women randomly assigned to intervention group
  Interventions: Other: Knowing your body; Behavioral: Healthy Lifestyle

INTERVENTIONS:
Other: Knowing your body — Women will receive the "Knowing your body" kit. The kit contains: 6 ovulation test strips, a 12 month menstrual log sheet/calendar, and a thermometer to help women determine their body temperature; and educational materials that contain information on female body parts involved in pregnancy, hormones and the menstrual cycle, how birth control works, body temperature changes, characteristics of cervical fluid, and adapting to pregnancy during the first trimester. Participants will receive a total of 10 visits. During the first visit, the nursing student/community health workers team will review the intervention kit and continue to discuss topics related to women's health during subsequent visits.
  Arms: Knowing your body
Behavioral: Healthy Lifestyle — Women will receive educational materials on healthy lifestyle such as maintaining good nutrition and the importance of folic acid for women of childbearing age during the first visit. Participants will receive a total of 10 visits. The nursing student/community health workers team will continue to discuss topics related to promoting healthy lifestyle during subsequent visits.

SUMMARY:
This study examines the efficacy of the "Preconception Reproductive Knowledge Promotion (PREKNOP)" intervention, designed to promote women's reproductive health and positive pregnancy outcomes. The study's goal is to educate low-income women about reproductive changes related to their menstrual cycle. The main hypothesis of the study is that women who receive the PREKNOP intervention will report reduced risk of unplanned pregnancy and increased reproductive knowledge, self-efficacy about that knowledge, and pregnancy planning ability.

DETAILED DESCRIPTION:
This study is a randomized, controlled trial of the PREKNOP intervention in a sample of 120 women 18-44 years old. Teams of nursing students and community health workers will administer the 12-month intervention. In addition to 10 home visits during which women will receive information on the female reproductive system and the expected monthly cyclical changes, PREKNOP will consist of use of ovulation test kits, a 12-month menstrual calendar, a digital thermometer, and educational brochures covering: the female reproductive anatomy, hormones and menstrual cycle, how to recognize ovulation period, various methods of birth control and how they work, and early pregnancy symptoms.

ELIGIBILITY:
Inclusion Criteria:

* low-income women of childbearing age

Exclusion Criteria:

* Menopause
* Hysterectomy

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-02; Primary Completion 2017-04-30 (Estimated); Study Completion 2017-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline reproductive knowledge of ovulation, menstrual cycle, peak fertile times, and early signs of pregnancy. | Baseline, 3, 6, 12, 18 and 24 months
  The investigators will measure if there is an increase in reproductive knowledge of ovulation time, menstrual cycle, peak fertile times, and early signs of pregnancy among the 120 participants in the study. The investigators will compare if there is higher increase in knowledge among the intervention group compared to the 60 participants in control group.

SECONDARY OUTCOMES:
Change from baseline number of unplanned pregnancies | Baseline, 3 months, 6 months, 12 months, 18months, 24 months
  The investigators will measure if there is a change in the number of unplanned pregnancies among the intervention group compared to the control group.

OTHER OUTCOMES:
Change in self-efficacy about reproductive knowledge and pregnancy planning ability | Baseline, 3 months, 6 months, 12 months, 18 months, 24 months
  The investigators will measure if there is an increase in self-efficacy score among the 120 participants in the study. The investigators will compare if there is higher increase among the 60 participants in the intervention group compared to the 60 participants in the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Adejoke B Ayoola, RN, PhD, Principal Investigator — Calvin College
Locations (1):
- Calvin College Nursing Department Community sites, Grand Rapids, Michigan, United States

REFERENCES:
- [Background] Ayoola AB, Nettleman M, Brewer J. Reasons for unprotected intercourse in adult women. J Womens Health (Larchmt). 2007 Apr;16(3):302-10. doi: 10.1089/jwh.2007.0210. PMID 17439376
- [Background] Nettleman MD, Chung H, Brewer J, Ayoola A, Reed PL. Reasons for unprotected intercourse: analysis of the PRAMS survey. Contraception. 2007 May;75(5):361-6. doi: 10.1016/j.contraception.2007.01.011. Epub 2007 Mar 12. PMID 17434017
- [Background] Finer LB, Zolna MR. Unintended pregnancy in the United States: incidence and disparities, 2006. Contraception. 2011 Nov;84(5):478-85. doi: 10.1016/j.contraception.2011.07.013. Epub 2011 Aug 24. PMID 22018121
- [Background] Dott M, Rasmussen SA, Hogue CJ, Reefhuis J; National Birth Defects Prevention Study. Association between pregnancy intention and reproductive-health related behaviors before and after pregnancy recognition, National Birth Defects Prevention Study, 1997-2002. Matern Child Health J. 2010 May;14(3):373-81. doi: 10.1007/s10995-009-0458-1. Epub 2009 Feb 28. PMID 19252975
- [Background] Ayoola AB, Zandee GL, Johnson E, Pennings K. Contraceptive use among low-income women living in medically underserved neighborhoods. J Obstet Gynecol Neonatal Nurs. 2014 Jul-Aug;43(4):455-64. doi: 10.1111/1552-6909.12462. Epub 2014 Jun 24. PMID 24958447
- [Background] Ayoola AB, Zandee GL. Low-income women's recommendations for promoting early pregnancy recognition. J Midwifery Womens Health. 2013 Jul-Aug;58(4):416-22. doi: 10.1111/jmwh.12078. Epub 2013 Jul 23. PMID 23879232